CLINICAL TRIAL: NCT04318535
Title: An Open Label, Randomized, Balanced, Three Treatment, Three Period, Three Sequence, Single Dose, Crossover Study to Evaluate the Bioequivalence of Test Griseofulvin Tablets, 500 mg Versus Reference Griseofulvin Tablets, 500 mg as Well as Dose Proportionality of Test Griseofulvin Tablets, 250 mg and 500 mg, in Healthy, Adult Participants Under Fed Conditions
Brief Title: Bioequivalence (BE) Study of Test Griseofulvin 500 Milligram (mg) Tablets Versus Reference and Dose Proportionality Study of Test Griseofulvin 250 mg and 500 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 212504
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Results first posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-11

CONDITIONS: Antifungal Agents
Keywords: Griseofulvin; Bioequivalence; Dose proportionality; Dermatophytosis
MeSH Terms: conditions — Tinea | interventions — Griseofulvin

STUDY DESIGN:
Intervention Model Description: The whole study will be divided into three treatment periods. For each treatment period, eligible participants will be randomized to either T1T2R, T2RT1 or RT1T2 treatment sequence according to 1:1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Participants receiving T1T2R (Experimental): Participants will receive a single oral dose of Griseofulvin T1: 1 x 500 mg Tablet once in Period 1 on Day 1 followed by a washout period of at least 7 days. In Period 2 on Day 8, same participants will receive Griseofulvin T2: 1 x 250 mg Tablet once followed by a washout period of at least 7 days. In Period 3 on Day 15, same participants will receive Griseofulvin R: 1 x 500 mg Tablet once. All the above-mentioned doses will be administered with 240 +- 2 milliliters (mL) of water at ambient temperature under fed condition.
  Interventions: Drug: Griseofulvin 500 mg; Drug: Griseofulvin 250 mg; Drug: Reference Griseofulvin 500 mg
- Participants receiving T2RT1 (Experimental): Participants will receive a single oral dose of Griseofulvin T2: 1 x 250 mg Tablet once in Period 1 on Day 1 followed by a washout period of at least 7 days. In Period 2 on Day 8, same participants will receive Griseofulvin R: 1 x 500 mg Tablet once followed by a washout period of at least 7 days. In Period 3 on Day 15, same participants will receive Griseofulvin T1: 1 x 500 mg Tablet once. All the above-mentioned doses will be administered with 240 +- 2 milliliters (mL) of water at ambient temperature under fed condition.
  Interventions: Drug: Griseofulvin 500 mg; Drug: Griseofulvin 250 mg; Drug: Reference Griseofulvin 500 mg
- Participants receiving RT1T2 (Experimental): Participants will receive a single oral dose of Griseofulvin R: 1 x 500 mg Tablet once in Period 1 on Day 1 followed by a washout period of at least 7 days. In Period 2 on Day 8, same participants will receive Griseofulvin T1: 1 x 500 mg Tablet once followed by a washout period of at least 7 days. In Period 3 on Day 15, same participants will receive Griseofulvin T2: 1 x 250 mg Tablet once. All the above-mentioned doses will be administered with 240 +- 2 milliliters (mL) of water at ambient temperature under fed condition.
  Interventions: Drug: Griseofulvin 500 mg; Drug: Griseofulvin 250 mg; Drug: Reference Griseofulvin 500 mg

INTERVENTIONS:
Drug: Griseofulvin 500 mg — Griseofulvin 500 mg will be administered as an oral tablet once in each treatment period under fed condition.
Drug: Griseofulvin 250 mg — Griseofulvin 250 mg will be administered as an oral tablet once in each treatment period under fed condition.
Drug: Reference Griseofulvin 500 mg — Reference Griseofulvin 500 mg will be administered as an oral tablet once in each treatment period under fed condition.

SUMMARY:
Griseofulvin is an antifungal agent used in treatment of Dermatophytosis caused by Microsporum spp. (species), Trichophyton spp., Epidermophyton spp., where topical therapy is considered inappropriate or has failed. Approved dose of Griseofulvin in Adults (greater than or equal to 50 kg) in India is 500 to 1,000 mg daily, but not less than 10 mg/kg bodyweight daily. As per the World health organization (WHO) guidance, Griseofulvin belongs to Biopharmaceutical Classification System (BCS) Class 2 ("low" solubility-"high" permeability). A Bioequivalence (BE) study will be conducted in India to estimate in vivo behavior (Pharmacokinetic characteristics) of Griseofulvin 500 tablets and dose proportionality study for Griseofulvin 250 mg and 500 mg tablets. This is an open label, randomized, balanced, three treatment period, three sequence, single dose, crossover study that will evaluate the bioequivalence of Griseofulvin tablets 500 mg test product (T1) versus Griseofulvin tablets 500 mg reference product (R) as well as dose proportionality of Griseofulvin tablets 250 mg test product (T2) with Griseofulvin tablets 500 mg T1 in healthy, adult participants under fed conditions. Eligible participants enrolled will be randomized to either of the three treatment sequence periods, T1T2R, T2RT1 or RT1T2 according to 1:1:1 ratio. The total duration of clinical phase will be approximately 20 days from Day-1 to Day 19 including a washout period of at least 7 days (not more than 14 days) for each treatment period. A total of 36 healthy, adult participants will be enrolled in this study and the above mentioned doses of Griseofulvin will be administered under fed conditions. Participants will be followed up 5 days after last dosing.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 45 years of age inclusive, at the time of signing the informed consent.
* Participants who are healthy as determined by the investigator or medically qualified designee on a medical evaluation including medical baseline history, physical examination and vital sign examination (blood pressure, pulse rate, respiration rate and body temperature).
* Participants with clinically acceptable findings as determined by hematology, biochemistry, urinalysis, 12 lead electrocardiogram (ECG).
* Participant's willingness to follow the protocol requirements especially abstaining from xanthine containing food or beverages (chocolates, tea, coffee or cola drinks) or grapefruit or grapefruit juice, any alcoholic products, the use of cigarettes and the use of tobacco products from 48 hours before the start of dosing until after collection of the final pharmacokinetic sample and adherence to food, fluid and posture restrictions.
* Participants with no history of significant alcoholism (Volunteers who do not have habit of heavy drinking which is defined as regular intake of more than 2 units of alcohol per day for male and 1 unit for female [I unit= 150 mL of wine or 360 mL of beer or 45 mL of 40 percent (%) of alcohol]).
* Participants with no history of drug abuse (benzodiazepines and barbiturates) for the last one month and other illegal drugs for the last 6 months.
* Participants who are non-smokers and ex-smokers will be included. "Ex-smokers are someone who completely stopped smoking for at least 3 months."
* Body mass index (BMI) within the range 18.5-30 kilogram per meter square (kg/m^2) (inclusive) and weight >= 50 kg.
* Healthy Male and non-pregnant female: Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Male participants are eligible to participate if they agree to the following during the treatment period and for at least six months after the last dose of study treatment.

  • Refrain from donating sperm as well as agree to use contraception/barrier as detailed below
  1. Agree to use a male condom and should also be advised for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.
  2. Agree to use male condom when engaging in any activity that allows for passage of ejaculate to another person.
* A female participant is eligible to participate if she is not pregnant and intending to become pregnant or breastfeeding, and at least one of the following conditions applies:

  * Is not a woman of childbearing potential (WOCBP) OR
  * Is a WOCBP and using a contraceptive method that is highly effective, with a failure rate of <1% during the treatment period and for at least 1 month after the last dose of study treatment. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study treatment.
  * A WOCBP must have a negative highly sensitive pregnancy test (serum as required by local regulations) within 1 day before each dose of study treatment (The participant must be excluded from participation if the serum pregnancy result is positive).

    b) Additional requirements for pregnancy testing during and after study treatment.

    c) The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Known history of hypersensitivity to Griseofulvin.
* Participants who have taken prescription medications or over-the-counter products (including vitamins, minerals and/or herbal supplements) within 14 days prior to administration of Investigational Medicinal Product (IMP).
* Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract, blood-forming organs, etc.
* History of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic, hematological, gastrointestinal, endocrine, immunological or psychiatric diseases.
* History of malignancy (including skin cancers) or other serious diseases.
* History of porphyria.
* Known history of Systemic lupus erythematosus (SLE) in the exclusion criteria.
* Participants consuming aspirin, oral contraceptive pills, phenobarbital, and warfarin having potential to trigger drug interactions with Griseofulvin for any ailment in the previous 28 days, prior to dosing day.
* Participation in a clinical drug study or bioequivalence study 90 days prior to period I dosing of the present study.
* Participants with positive Human Immuno Deficiency Virus (HIV) tests, Hepatitis B Surface Antigen (HBsAg) or Hepatitis-C tests.
* Found positive in breath alcohol test.
* Found positive in urine test for drug abuse.
* Blood donation 90 days prior to period I dosing of the present study.
* History of problem in swallowing pills.
* Any contraindication to blood sampling i.e. keloid formation.
* Sensitivity to heparin or heparin-induced thrombocytopenia.
* Premenarchal female participants.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Navi Mumbai, India

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label, randomized,3-treatment,3-period, single dose, crossover study. Bioequivalence between test Griseofulvin tablets (500 milligram [mg]) versus reference Griseofulvin tablets 500 mg and dose proportionality between test Griseofulvin tablets (250 mg and 500 mg) were evaluated in healthy adult participants under fed conditions.
Pre-assignment Details: A total of 36 participants were enrolled and received study treatment. The study had 3 periods: Period 1 (Day -1 to Day 5), Period 2 (Day 7 to Day 12) and Period 3 (Day 17 to Day 22) with a washout of atleast 7 days (not more than 14 days) between two subsequent dosing days.
Groups:
- Griseofulvin 500-T1/Griseofulvin 250-T2/Griseofulvin 500-R: Participants received a single oral dose of Griseofulvin 500 mg (Treatment 1 [T1]) in treatment period 1 (Day 1) followed by Griseofulvin 250 mg (T2) in treatment period 2 (Day 8) followed by Griseofulvin 500 mg (Reference [R]) in treatment period 3 (Day 18). There was a washout period of at least 7 days between 2 subsequent dosing days.
- Griseofulvin 250-T2/Griseofulvin 500-R/Griseofulvin 500-T1: Participants received a single oral dose of Griseofulvin 250 mg (T2) in treatment period 1 (Day 1) followed by Griseofulvin 500 mg (R) in treatment period 2 (Day 8) followed by Griseofulvin 500 mg (T1) in treatment period 3 (Day 18). There was a washout period of at least 7 days between 2 subsequent dosing days.
- Griseofulvin 500-R/Griseofulvin 500-T1/Griseofulvin 250-T2: Participants received a single oral dose of Griseofulvin 500 mg (R) in treatment period 1 (Day 1) followed by Griseofulvin 500 mg (T1) in treatment period 2 (Day 8) followed by Griseofulvin 250 mg (T2) in treatment period 3 (Day 18). There was a washout period of at least 7 days between 2 subsequent dosing days.
Period: Treatment Period 1 (Day -1 to Day 5)
Arm/Group | Griseofulvin 500-T1/Griseofulvin 250-T2/Griseofulvin 500-R | Griseofulvin 250-T2/Griseofulvin 500-R/Griseofulvin 500-T1 | Griseofulvin 500-R/Griseofulvin 500-T1/Griseofulvin 250-T2
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0
Period: Period1washout(Atleast 7 Days Post-dose)
Arm/Group | Griseofulvin 500-T1/Griseofulvin 250-T2/Griseofulvin 500-R | Griseofulvin 250-T2/Griseofulvin 500-R/Griseofulvin 500-T1 | Griseofulvin 500-R/Griseofulvin 500-T1/Griseofulvin 250-T2
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0
Period: Treatment Period 2 (Day 7 to Day 12)
Arm/Group | Griseofulvin 500-T1/Griseofulvin 250-T2/Griseofulvin 500-R | Griseofulvin 250-T2/Griseofulvin 500-R/Griseofulvin 500-T1 | Griseofulvin 500-R/Griseofulvin 500-T1/Griseofulvin 250-T2
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0
Period: Period2washout(Atleast 7 Days Post-dose)
Arm/Group | Griseofulvin 500-T1/Griseofulvin 250-T2/Griseofulvin 500-R | Griseofulvin 250-T2/Griseofulvin 500-R/Griseofulvin 500-T1 | Griseofulvin 500-R/Griseofulvin 500-T1/Griseofulvin 250-T2
Started | 12 | 12 | 12
Completed | 12 | 11 | 12
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Period: Treatment Period 3 (Day 17 to Day 22)
Arm/Group | Griseofulvin 500-T1/Griseofulvin 250-T2/Griseofulvin 500-R | Griseofulvin 250-T2/Griseofulvin 500-R/Griseofulvin 500-T1 | Griseofulvin 500-R/Griseofulvin 500-T1/Griseofulvin 250-T2
Started | 12 | 11 | 12
Completed | 12 | 11 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Treated Participants: All participants received a single oral dose of Griseofulvin 500 mg tablet (T1), Griseofulvin 250 mg tablet (T2) and Griseofulvin 500 mg tablet (R) in either Period 1 or Period 2 or Period 3 as per randomization schedule.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.08 (5.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - South East Asian Heritage | 36

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) for Griseofulvin
Description: Blood samples were collected to measure Cmax at indicated time-points. Pharmacokinetic parameters were measured using standard non-compartmental methods. For Griseofulvin 250 mg (T2), dose-normalized Cmax (observed value multiplied by 2) is reported. Adjusted geometric mean and standard error have been presented for all treatments. Adjusted geometric mean is the antilog (exponential) of the least squares mean of the log-transformed data. Statistical analysis of pharmacokinetic parameters was done using mixed model for evaluation of bioquivalence. Point estimate and 90% confidence interval for the ratio of geometric least square mean of the test Griseofulvin 500 mg (T1) to the reference Griseofulvin 500 mg (R) were calculated for Cmax to assess bioequivalence.
Time Frame: Pre-dose (within 1 hour prior to dosing) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 24, 48, 72 and 96 hours post-dose in each period
Population: Bioequivalence (BE) Analysis Set Population comprised of participants completing at least 2 periods with 500 mg test and 500 mg reference treatments of the study. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Standard Error); unit: Nanograms per milliliter
Groups:
- Griseofulvin 500 mg (T1): All participants received a single oral dose of Griseofulvin 500 mg tablet (T1) in either Period 1 or Period 2 or Period 3 as per randomization schedule.
- Griseofulvin 250 mg (T2): All participants received a single oral dose of Griseofulvin 250 mg tablet (T2) in either Period 1 or Period 2 or Period 3 as per randomization schedule.
- Griseofulvin 500 mg (R): All participants received a single oral dose of Griseofulvin 500 mg tablet (R) in either Period 1 or Period 2 or Period 3 as per randomization schedule.
Arm/Group | Griseofulvin 500 mg (T1) | Griseofulvin 250 mg (T2) | Griseofulvin 500 mg (R)
Number analyzed (Participants) | 35 | 35 | 35
Nanograms per milliliter | 2229 (0.03262) | 2877 (0.03457) | 1927 (0.03262)
Statistical Analysis 1: Comparison: Griseofulvin 500 mg (T1) vs Griseofulvin 500 mg (R); Test type: Equivalence — Bioequivalence was to be determined if the 90% confidence interval of the geometric least square mean ratio of Cmax falls within the 0.80-1.25 range; Ratio of geometric least square mean = 1.157, 90% CI 2-sided [1.103 to 1.213] — T1 versus R was the primary interest of comparison for this outcome measure

2. Primary Outcome: Area Under Plasma Concentration-time Curve (AUC) From Zero Hours to Time of Last Quantifiable Concentration (AUC[0-t]) for Griseofulvin
Description: Blood samples were collected to measure AUC(0-t) at indicated time-points. Pharmacokinetic parameters were measured using standard non-compartmental methods. For Griseofulvin 250 mg (T2), dose-normalized AUC(0-t) (observed value multiplied by 2) is reported. Adjusted geometric mean and standard error have been presented for all treatments. Adjusted geometric mean is the antilog (exponential) of the least squares mean of the log-transformed data. Statistical analysis of pharmacokinetic parameters was done using mixed model for evaluation of bioquivalence. Point estimate and 90% confidence interval for the ratio of geometric least square mean of the test Griseofulvin 500 mg (T1) to the reference Griseofulvin 500 mg (R) were calculated for AUC(0-t) to assess bioequivalence.
Time Frame: as for outcome 1
Population: Bioequivalence (BE) Analysis Set Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Standard Error); unit: Hours*nanogram per milliliter
Arm/Group | Griseofulvin 500 mg (T1) | Griseofulvin 250 mg (T2) | Griseofulvin 500 mg (R)
Number analyzed (Participants) | 35 | 35 | 35
Hours*nanogram per milliliter | 54993 (0.05305) | 66788 (0.05560) | 53274 (0.05305)
Statistical Analysis 1: Comparison: Griseofulvin 500 mg (T1) vs Griseofulvin 500 mg (R); Test type: Equivalence — Bioequivalence was to be determined if the 90% confidence interval of the geometric least square mean ratio of AUC(0-t) falls within the 0.80-1.25 range; Ratio of geometric least square mean = 1.032, 90% CI 2-sided [0.974 to 1.094] — T1 versus R was the primary interest of comparison for this outcome measure

3. Primary Outcome: AUC From Time Zero Extrapolated to Infinity (AUC[0-inf]) for Griseofulvin
Description: Blood samples were collected to measure AUC(0-inf) at indicated time-points. Pharmacokinetic parameters were measured using standard non-compartmental methods. For Griseofulvin 250 mg (T2), dose-normalized AUC(0-inf) (observed value multiplied by 2) is reported. Adjusted geometric mean and standard error have been presented for all treatments. Adjusted geometric mean is the antilog (exponential) of the least squares mean of the log-transformed data. Statistical analysis of pharmacokinetic parameters was done using mixed model for evaluation of bioquivalence. Point estimate and 90% confidence interval for the ratio of geometric least square mean of the test Griseofulvin 500 mg (T1) to the reference Griseofulvin 500 mg (R) were calculated for AUC(0-inf) to assess bioequivalence.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Standard Error); unit: Hours*nanogram per milliliter
Arm/Group | Griseofulvin 500 mg (T1) | Griseofulvin 250 mg (T2) | Griseofulvin 500 mg (R)
Number analyzed (Participants) | 35 | 35 | 35
Hours*nanogram per milliliter | 56746 (0.05460) | 69564 (0.05630) | 55100 (0.05460)
Statistical Analysis 1: Comparison: Griseofulvin 500 mg (T1) vs Griseofulvin 500 mg (R); Test type: Equivalence — Bioequivalence was to be determined if the 90% confidence interval of the geometric least square mean ratio of AUC(0-inf) falls within the 0.80-1.25 range; Ratio of geometric least square mean = 1.030, 90% CI 2-sided [0.971 to 1.093] — T1 versus R was the primary interest of comparison for this outcome measure

4. Primary Outcome: Dose Proportionality of Griseofulvin Using AUC(0-t) Following a Single Dose
Description: Blood samples were collected at indicated time-points for pharmacokinetic analysis. Pharmacokinetic parameters were measured using standard non-compartmental methods. Dose proportionality was assessed using mixed model. Slope and 90% confidence interval for the slope are presented. For Griseofulvin 250 mg (T2), dose-normalized (observed value multiplied by 2) AUC(0-t) was used during calculation of dose proportionality.
Time Frame: as for outcome 1
Population: Dose Proportionality Analysis Set Population comprised of participants completing at least 2 periods with 500 mg test (T1) and 250 mg test (T2) treatments of the study. Only those participants with data available at the specified time points were analyzed.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Groups:
- Griseofulvin 250 mg to 500 mg: All participants received a single oral dose of Griseofulvin 250 mg or 500 mg tablet in either Period 1 or Period 2 or Period 3 as per randomization schedule.
Arm/Group | Griseofulvin 250 mg to 500 mg
Number analyzed (Participants) | 35
Slope of log dose | 1.214 [1.156 to 1.275]

5. Primary Outcome: Dose Proportionality of Griseofulvin Using Cmax Following a Single Dose
Description: Blood samples were collected at indicated time-points for pharmacokinetic analysis. Pharmacokinetic parameters were measured using standard non-compartmental methods. Dose proportionality was assessed using mixed model. Slope and 90% confidence interval for the slope are presented. For Griseofulvin 250 mg (T2), dose-normalized (observed value multiplied by 2) Cmax was used during calculation of dose proportionality.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | Griseofulvin 250 mg to 500 mg
Number analyzed (Participants) | 35
Slope of log dose | 1.290 [1.239 to 1.344]

6. Secondary Outcome: Number of Participants With Any Serious Adverse Event (SAE) and Any Non-serious Adverse Event (Non-SAE)
Description: An adverse event was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the medicinal product. An SAE was any untoward medical occurrence resulting in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, congenital anomaly/birth defect or any other other important medical event that may jeopardize the participant or may require medical or surgical treatment to prevent one of the other outcomes listed before.
Time Frame: Up to Day 22
Population: Safety Analysis Set Population comprised of all randomized participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Griseofulvin 500 mg (T1) | Griseofulvin 250 mg (T2) | Griseofulvin 500 mg (R)
Number analyzed (Participants) | 36 | 36 | 36
Participants
  Any SAE | 0 | 0 | 0
  Any non-SAE | 0 | 0 | 1

7. Secondary Outcome: Number of Participants With Any Abnormality in Vital Signs
Description: Systolic blood pressure (SBP), diastolic blood pressure (DBP), pulse rate, respiration rate and body temperature were measured in semi-supine position after 5 minutes rest. The clinically acceptable range included; SBP: 85 millimeters of mercury (mmHg) to 160 mmHg; DBP: 45 mmHg to 100 mmHg; pulse rate: 40 beats per minute to 110 beats per minute; respiration rate: 8 breaths per minute to 20 breaths per minute; body temperature: 35.5 degrees Celsius to 37.8 degrees Celsius. Number of participants with any abnormality in vital signs are presented.
Time Frame: Up to Day 22
Population: Safety Analysis Set Population
Measure: Count of Participants; unit: Participants
Arm/Group | Griseofulvin 500 mg (T1) | Griseofulvin 250 mg (T2) | Griseofulvin 500 mg (R)
Number analyzed (Participants) | 36 | 36 | 36
Participants
  SBP | 0 | 0 | 0
  DBP | 0 | 0 | 0
  Pulse rate | 0 | 0 | 0
  Respiration rate | 0 | 0 | 0
  Body temperature | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Any Abnormality in Hematology Parameters
Description: Blood samples were collected at indicated time points for assessment of hematology parameters. The clinically acceptable range included; hemoglobin: 12.3-18.0 grams per deciliter (g/dL) (for male) and 11.0-16.0 g/dL (for female), erythrocyte count: 4.0-7.1*10^12 cells per liter (for male) and 3.6-5.6*10^12 cells per liter (for female), hematocrit: 0.41-0.50 proportion of red blood cells in blood (Male) and 0.35-0.44 proportion of red blood cells in blood (Female), Mean Corpuscular Volume (MCV): 80-96 femtoliters, Mean Corpuscular Hemoglobin (MCH): 27.5-33.2 picogram , Mean Corpuscular Hemoglobin Concentration (MCHC): 33.4-35.5 g/dL, White Blood Cell (WBC) count: 3960-12100 cells per microliter, platelet count: 135-495*10^9 cells per liter, neutrophils: 36-88%, eosinophils: up to 14%, basophils: 0-2%, lymphocytes: 18-44%, monocytes: 2-10% of total cells. Number of participants with any abnormality in hematology parameters are presented.
Time Frame: Up to Day 22
Population: Safety Analysis Set Population
Measure: Count of Participants; unit: Participants
Arm/Group | Griseofulvin 500 mg (T1) | Griseofulvin 250 mg (T2) | Griseofulvin 500 mg (R)
Number analyzed (Participants) | 36 | 36 | 36
Participants
  Hemoglobin | 0 | 0 | 0
  Erythrocyte count | 0 | 0 | 0
  Hematocrit | 0 | 0 | 0
  MCV | 0 | 0 | 0
  MCH | 0 | 0 | 0
  MCHC | 0 | 0 | 0
  WBC count | 0 | 0 | 1
  Neutrophils count | 0 | 0 | 0
  Eosinophils count | 0 | 0 | 0
  Basophils count | 0 | 0 | 0
  Lymphocytes count | 0 | 0 | 0
  Monocytes count | 0 | 0 | 0
  Platelet count | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Any Abnormality in Clinical Chemistry Parameters
Description: Blood samples were collected at indicated time points for assessment of clinical chemistry parameters. The clinically acceptable range included; blood urea: Up to 55 milligrams per deciliter (mg/dL), random blood glucose: 63-140 mg/dL, blood urea nitrogen: Up to 25 mg/dL, serum creatinine: 0.6-1.3 mg/dL (Male) and 0.4-1.0 mg/dL (Female), total serum bilirubin: 0.00-1.47 mg/dL, direct serum bilirubin: 0.0-0.3 mg/dL, indirect serum bilirubin: 0.0-1.5 mg/dL, aspartate aminotransferase (AST): Up to 70 units per liter (U/L) (Male) and Up to 50 U/L (Female). Number of participants with any abnormality in clinical chemistry parameters are presented.
Time Frame: Up to Day 22
Population: Safety Analysis Set Population
Measure: Count of Participants; unit: Participants
Arm/Group | Griseofulvin 500 mg (T1) | Griseofulvin 250 mg (T2) | Griseofulvin 500 mg (R)
Number analyzed (Participants) | 36 | 36 | 36
Participants
  Blood urea | 0 | 0 | 0
  Random blood glucose | 0 | 0 | 0
  Blood urea nitrogen | 0 | 0 | 0
  Serum creatinine | 0 | 0 | 0
  Total serum bilirubin | 0 | 0 | 0
  Direct serum bilirubin | 0 | 0 | 0
  Indirect serum bilirubin | 0 | 0 | 0
  AST | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Any Abnormality in Clinical Chemistry Parameter: Alanine Aminotransferase (ALT)
Description: Blood samples were collected at indicated time points for assessment of clinical chemistry parameter. The clinically acceptable range for ALT included; Up to 7270 units per liter (U/L) (Male) and Up to 50 U/L (Female). Number of participants with any abnormality in ALT levels are presented.
Time Frame: Days -1, 7, 17 and 22
Population: Safety Analysis Set Population
Measure: Count of Participants; unit: Participants
Arm/Group | Griseofulvin 500 mg (T1) | Griseofulvin 250 mg (T2) | Griseofulvin 500 mg (R)
Number analyzed (Participants) | 36 | 36 | 36
Participants
  Day -1 | 0 | 0 | 0
  Day 7 | 0 | 0 | 0
  Day 17 | 0 | 0 | 0
  Day 22 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Positive Results in Serum Beta-human Chorionic Gonadotropin (Beta-hCG) Level (Females Participants)
Description: Blood samples were collected at indicated time points for assessment of serum beta-hCG (serum pregnancy test) for female participants. Number of participants with positive results in serum beta-hCG levels are presented.
Time Frame: Days -1, 7, 17 and 22
Population: Safety Analysis Set Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Griseofulvin 500 mg (T1) | Griseofulvin 250 mg (T2) | Griseofulvin 500 mg (R)
Number analyzed (Participants) | 5 | 5 | 5
Participants
  Day -1 | 0 | 0 | 0
  Day 7 | 0 | 0 | 0
  Day 17 | 0 | 0 | 0
  Day 22 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Abnormal Urinalysis Dipstick Results
Description: Urine samples were collected to assess glucose, ketones, occult blood, protein, urobilinogen and bilirubin by dipstick method. The dipstick test gave results in a semi-quantitative manner, and results can be read as Negative, Trace, 1+, 2+ indicating proportional concentrations in the urine sample. Clinically acceptable range included 'negative' and 'trace' results. Number of participants with any abnormal urinalysis parameters are presented.
Time Frame: Up to Day 22
Population: Safety Analysis Set Population
Measure: Count of Participants; unit: Participants
Arm/Group | Griseofulvin 500 mg (T1) | Griseofulvin 250 mg (T2) | Griseofulvin 500 mg (R)
Number analyzed (Participants) | 36 | 36 | 36
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were reported from start of study treatment (Day 1) up to Day 22
Description: Non-SAEs and SAEs were reported for Safety Analysis Set Population. Adverse events were presented treatment-wise.
Arm/Group | Griseofulvin 500 mg (T1) | Griseofulvin 250 mg (T2) | Griseofulvin 500 mg (R)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 1/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Griseofulvin 500 mg (T1) (N=36) | Griseofulvin 250 mg (T2) (N=36) | Griseofulvin 500 mg (R) (N=36)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT04318535/SAP_000.pdf
  • Study Protocol (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/35/NCT04318535/Prot_001.pdf